CLINICAL TRIAL: NCT01718483
Title: The SPD489-343, Phase 3, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Dose-optimization Study to Evaluate the Efficacy, Safety, and Tolerability of SPD489 in Adults Aged 18-55 Years With Moderate to Severe Binge Eating Disorder
Brief Title: SPD489 in Adults Aged 18-55 Years With Moderate to Severe Binge Eating Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD489-343; 2012-003309-91 (EudraCT Number)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPD489 (Lisdexamfetamine dimesylate) (Experimental)
  Interventions: Drug: SPD489 (Lisdexamfetamine dimesylate)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD489 (Lisdexamfetamine dimesylate) — 50 or 70 mg administered orally, once-daily for up to 12 weeks
  Other Names: Vyvanse, Venvanse, LDX
  Arms: SPD489 (Lisdexamfetamine dimesylate)
Drug: Placebo — Administered once-daily, orally, for up to 12 weeks
  Arms: Placebo

SUMMARY:
The primary objective of the study is to demonstrate the efficacy of SPD489 compared with placebo in adults (18 55 years of age inclusive) with moderate to severe Binge Eating Disorder at Visit 8 (Weeks 11 and 12) as measured by the number of binge days (defined as days during which at least 1 binge episode occurs) per week as assessed by clinical interview based on subject diary

ELIGIBILITY:
Inclusion Criteria -

1. Subject is between 18-55 years of age.
2. Subject meets the following DSM-IV-TR criteria for a diagnosis of BED:

   Recurrent episodes of binge eating. An episode of binge eating is characterized by both of the following: eating, in a discrete period of time (eg, within a 2-hour period) an amount of food that is definitely larger than most people would eat in a similar period of time under similar conditions, and a sense of lack of control over the eating (eg, a feeling that one cannot stop eating or control what or how much one is eating).

   The binge eating episodes are associated with at least 3 of the following: eating much more rapidly than normal; eating until uncomfortably full; eating large amounts of food when not feeling physically hungry; eating alone because of being embarrassed by how much one is eating; feeling disgusted with oneself, depressed, or feeling very guilty after overeating.

   Marked distress regarding binge eating. The binge eating occurs, on average, at least 2 days a week for 6 months. The episodes of binge eating do not occur exclusively during the course of bulimia nervosa or anorexia nervosa.
3. Subject's BED is of at least moderate severity with subjects reporting at least 3 binge eating days per week for the 14 days prior to the Baseline Visit (Visit 0) as documented in the subject's binge diary. A binge day is a day during which at least 1 binge eating episode occurs.
4. Female subjects must have a negative serum B HCG pregnancy test and a negative urine pregnancy test.

Exclusion Criteria-

1. Subject has concurrent symptoms of bulimia nervosa or anorexia nervosa.
2. Subject is receiving psychotherapy (eg, supportive psychotherapy, cognitive behavior therapy, interpersonal therapy) or weight loss support (eg, Weight Watchers) for BED within 3 months.
3. Subject has used psychostimulants to facilitate fasting or dieting as a part of their BED within 6 months.
4. Subject has a lifetime history of psychosis, mania, hypomania, dementia, or ADHD.
5. Subject is considered a suicide risk in the opinion of the investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the investigator.
6. Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems.
7. Subject has recently initiated treatment with a lipid-lowering medication (within the past 3 months).
8. Subject has a history of moderate or severe hypertension.
9. Subject is female and pregnant or nursing.
10. Subjects who have had bariatric surgery, lap bands, duodenal stents, or other procedures for weight loss.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 383 (Actual)
Dates: Start 2012-11-26 (Actual); Primary Completion 2013-09-25 (Actual); Study Completion 2013-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (50):
- United States (43):
  - Birmingham Research Group, Birmingham, Alabama
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Trimed Clinical Trials, Corona, California
  - Pharmacology Research Institute, Encino, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pacific Research Partners, LLC, Oakland, California
  - Research Across America, Santa Ana, California
  - Western Affiliated Research Institute, Inc., Denver, Colorado
  - Gulfcoast Clinical Research, Fort Myers, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Fidelity Clinical Research, Inc., Lauderhill, Florida
  - Compass Research LLC, Leesburg, Florida
  - Scientific Clinical Research Inc., North Miami, Florida
  - Uptown Research Institute, Chicago, Illinois
  - Alexian Brothers Behavioral Health Hospital, Hoffman Estates, Illinois
  - AMR Baber Research, Inc., Naperville, Illinois
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Cypress Medical Research Center, LLC, Wichita, Kansas
  - McLean Hospital, Belmont, Massachusetts
  - St. Charles Psychiatric Associates/Midwest Research Group, Saint Charles, Missouri
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Pacific Research for Research and Evaluation, Albuquerque, New Mexico
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Community Research, Cincinnati, Ohio
  - Midwest Clinical Research Center, LLC, Dayton, Ohio
  - North Star Medical Research, Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - The Clinical Trials Center, LLC, Jenkintown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Radiant Research, Inc., Anderson, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Future Search Trials, Austin, Texas
  - Futuresearch Trials of Dallas, L.P., Dallas, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Radiant Research, Inc., Murray, Utah
  - Neuropsychiatric Associates, LLC, Woodstock, Vermont
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Alliance Research Group, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Dean Foundation for Health, Research and Educations, Inc., Middleton, Wisconsin
- Germany (3):
  - Ernovis GmbH, Berlin
  - Klinische Forschung Dresden GmbH, Dresden
  - Studienzentrum Nordwest, Gemeinschaftspraxis, Westerstede
- Hospital Universitario Infanta Leonor, Madrid, Spain
- Sweden (3):
  - Lakarmottagning Ekdahl & Kronberg, Malmo
  - Sophiahemmet, Stockholm
  - Stockholm Center for Eating Disorders, Stockholm

REFERENCES:
- [Result] McElroy SL, Hudson J, Ferreira-Cornwell MC, Radewonuk J, Whitaker T, Gasior M. Lisdexamfetamine Dimesylate for Adults with Moderate to Severe Binge Eating Disorder: Results of Two Pivotal Phase 3 Randomized Controlled Trials. Neuropsychopharmacology. 2016 Apr;41(5):1251-60. doi: 10.1038/npp.2015.275. Epub 2015 Sep 9. PMID 26346638
- [Derived] Robertson B, Wu J, Fant RV, Schnoll SH, McElroy SL. Assessment of Amphetamine Withdrawal Symptoms of Lisdexamfetamine Dimesylate Treatment for Adults With Binge-Eating Disorder. Prim Care Companion CNS Disord. 2020 Mar 26;22(2):19m02540. doi: 10.4088/PCC.19m02540. PMID 32237290
- [Derived] Kornstein SG, Bliss C, Kando J, Madhoo M. Clinical Characteristics and Treatment Response to Lisdexamfetamine Dimesylate Versus Placebo in Adults With Binge Eating Disorder: Analysis by Gender and Age. J Clin Psychiatry. 2019 Feb 26;80(2):18m12378. doi: 10.4088/JCP.18m12378. PMID 30817099
- [Derived] Sheehan DV, Gasior M, McElroy SL, Radewonuk J, Herman BK, Hudson J. Effects of Lisdexamfetamine Dimesylate on Functional Impairment Measured on the Sheehan Disability Scale in Adults With Moderate-to-severe Binge Eating Disorder: Results from Two Randomized, Placebo-controlled Trials. Innov Clin Neurosci. 2018 Jun 1;15(5-6):22-29. PMID 30013816
- [Derived] Citrome L, Kando JC, Bliss C. Relationships between clinical scales and binge eating days in adults with moderate to severe binge eating disorder in two Phase III studies. Neuropsychiatr Dis Treat. 2018 Feb 15;14:537-546. doi: 10.2147/NDT.S158395. eCollection 2018. PMID 29497297

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 12-Nov-2012 and 19-June-2013 and locations included medical clinics & research centers.
Groups:
- PLACEBO: Placebo matching SPD489 capsule administered orally, once-daily, for up to 12 weeks.
- SPD489: SPD489 capsule 30 (titration purpose only), 50 or 70 milligram (mg) administered orally, once-daily for up to 12 weeks once the optimal dose is reached.
Period: Overall Study
Arm/Group | PLACEBO | SPD489
Started | 191 | 192
Treated | 187 | 192
Completed | 157 | 158
Not Completed | 34 | 34
Not completed — Withdrawal by Subject | 14 | 12
Not completed — Adverse Event | 5 | 12
Not completed — Lost to Follow-up | 8 | 3
Not completed — Protocol Violation | 4 | 2
Not completed — Other | 1 | 4
Not completed — Pregnancy | 1 | 1
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set was used for Baseline Measures. The Safety Analysis Set was defined as all randomized participants who took at least 1 dose of investigational product and who had at least 1 post-baseline safety assessment completed. Four participants did not receive investigational product, therefore n=379.
Groups:
- PLACEBO: Placebo matching SPD489 capsule administered orally, once-daily for up to 12 weeks.
- SPD489: SPD489 capsule 30 (titration purpose only), 50 or 70 mg administered orally, once-daily for up to 12 weeks once the optimal dose is reached.
- Total: Total of all reporting groups
Arm/Group | PLACEBO | SPD489 | Total
Number analyzed (Participants) | 187 | 192 | 379
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.6 (10.21) | 38.5 (10.4) | 38.1 (10.3)
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 102 | 98 | 200
  >=40 years | 85 | 94 | 179
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 165 | 328
  Male | 24 | 27 | 51
Region of Enrollment [Count of Participants; unit: Participants]
  GERMANY | 2 | 1 | 3
  SPAIN | 5 | 5 | 10
  SWEDEN | 15 | 13 | 28
  UNITED STATES | 165 | 173 | 338

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Binge Days Per Week at Visit 8 (Weeks 11-12)
Description: Binge days defined as days during which at least 1 binge episode occurred. As assessed by clinical interview based on participant binge diary.
Time Frame: Baseline and Visit 8 (Weeks 11-12)
Population: The Full Analysis Set was defined as all randomized participants who took at least 1 dose of investigational product and who had 1 post-baseline primary efficacy assessment (number of binge days per week calculated for at least 1 week).
Measure: Least Squares Mean (Standard Error); unit: Binge days per week
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 184 | 190
Binge days per week | -2.51 (0.125) | -3.87 (0.124)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis; Least squares mean difference = -1.35, 95% CI 2-sided [-1.70 to -1.01]

2. Secondary Outcome: Percentage of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I) Scores
Description: CGI-I consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: Up to 12 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 184 | 190
percentage of participants | 47.3 [40.1 to 54.5] | 82.1 [76.7 to 87.6]
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Chi-squared

3. Secondary Outcome: Percentage of Participants With a 4-Week Cessation From Binge Eating
Description: 4-week cessation from binge eating is defined as no binge eating episodes for 28 consecutive days prior to the last study visit.
Time Frame: Up to 12 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 184 | 190
percentage of participants | 14.1 [9.1 to 19.2] | 40.0 [33.0 to 47.0]
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Chi-squared

4. Secondary Outcome: Percent Change From Baseline in Body Weight at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 184 | 190
percent change | 0.11 (0.295) | -6.25 (0.292)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis; Least squares mean difference = -6.35, 95% CI 2-sided [-7.17 to -5.54]

5. Secondary Outcome: Change From Baseline in Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating (Y-BOCS-BE) Total Score at Week 12
Description: The Y-BOCS-BE measures the obsession of binge-eating thoughts and compulsiveness of binge-eating behaviors. The scale is a clinician-rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms). Total scores range from 0 to 40. Reduction in total score indicates improvement.
Time Frame: Baseline and Week 12
Population: The Full Analysis Set was defined as all randomized participants who took at least 1 dose of investigational product and who had 1 post-baseline primary efficacy assessment (number of binge days per week calculated for at least 1 week). Not all participants had data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 183 | 188
units on a scale | -8.28 (0.550) | -15.68 (0.546)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis; Least squares mean difference = -7.40, 95% CI 2-sided [-8.93 to -5.88]

6. Secondary Outcome: Change From Baseline in Fasting Triglyceride Levels at Up to 12 Weeks
Time Frame: Baseline and Week 12/Early termination (ET)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 183 | 190
millimole per liter (mmol/L) | 0.122 (0.0405) | -0.077 (0.0393)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, ANCOVA; Least squares mean difference = -0.199, 95% CI 2-sided [-0.310 to -0.088]

7. Secondary Outcome: Change From Baseline In Fasting Total Cholesterol Levels at Up to 12 Weeks
Time Frame: Baseline and Week 12/ET
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 183 | 190
mmol/L | -0.094 (0.0435) | -0.305 (0.0422)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, ANCOVA; Least squares mean difference = -0.211, 95% CI 2-sided [-0.330 to -0.092]

8. Secondary Outcome: Change From Baseline in Hemoglobin A1c Levels at Up to 12 Weeks
Time Frame: Baseline and Week 12/ET
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Percent hemoglobin
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 181 | 189
Percent hemoglobin | 0.01 (0.016) | -0.02 (0.015)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p = 0.308, ANCOVA; Least squares mean difference = -0.02, 95% CI 2-sided [-0.07 to 0.02]

9. Secondary Outcome: Binge Eating Response
Description: Response is based on the reduction in the number of binge eating episodes. Percentage of participants with response was reported. Responses were categorized as follows: 1-week Cessation = 100% reduction in binge episodes during the preceding 7 days. Marked Reduction = 99% to 75% reduction during the time since the previous visit. Moderate Reduction = 74% to 50% reduction during the time since the previous visit. Negative to Minimal Reduction = <50% reduction during the time since the previous visit.
Time Frame: Week 12/ET
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 184 | 187
percentage of participants
  1-week cessation | 26.6 | 47.1
  Marked Reduction | 15.2 | 31.6
  Moderate Reduction | 17.9 | 11.8
  Negative to Minimal Reduction | 40.2 | 9.6
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity is not adjusted for this secondary efficacy endpoint in this study

10. Secondary Outcome: Change From Baseline in the Number of Binge Episodes Per Week at Visit 8 (Weeks 11-12)
Time Frame: Baseline and Visit 8 (Weeks 11-12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Binge episodes per week
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 184 | 190
Binge episodes per week | -3.49 (0.170) | -5.27 (0.168)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis — Multiplicity is not adjusted for this secondary efficacy endpoint in this study; Least squares mean difference = -1.77, 95% CI 2-sided [-2.24 to -1.30]

11. Secondary Outcome: Change From Baseline in Eating Inventory Scores at Week 12
Description: The Eating Inventory also known as the Three-Factor Eating Questionnaire is a 51-item self-reported questionnaire intended to assess 3 dimensions of eating behavior. There are 36 true/false items, 14 items on a 4-point Likert scale (1=eat rarely to 4=always), and 1 item on a 6-point Likert scale (1=eat whatever you want to 6=constantly limiting food intake). Cognitive Restraint score ranges from 0-21. Hunger score ranges from 0-14. Disinhibition score ranges from 0-16. Higher scores denote higher levels of restrained eating, disinhibited eating and predisposition to hunger.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 184 | 188
units on a scale
  Cognitive Restraint of Eating | 1.63 (0.331) | 3.27 (0.329)
  Disinhibition of Eating | -2.12 (0.286) | -6.31 (0.285)
  Perceived Hunger | -1.90 (0.286) | -6.60 (0.285)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Cognitive Restraint of Eating; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis — Multiplicity is not adjusted for this secondary efficacy endpoint in this study; Least squares mean difference = 1.65, 95% CI 2-sided [0.72 to 2.57]
Statistical Analysis 2: Comparison: PLACEBO vs SPD489; Disinhibition of Eating; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis — Multiplicity is not adjusted for this secondary efficacy endpoint in this study; Least squares mean difference = -4.19, 95% CI 2-sided [-4.98 to -3.39]
Statistical Analysis 3: Comparison: PLACEBO vs SPD489; Perceived Hunger; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis — Multiplicity is not adjusted for this secondary efficacy endpoint in this study; Least squares mean difference = -4.70, 95% CI 2-sided [-5.49 to -3.91]

12. Secondary Outcome: Change From Baseline in Binge Eating Scale (BES) Score at Week 12
Description: The BES is a self-reported questionnaire containing 16 items designed to assess behavioral, affective, and attitudinal components of the subjective experience of binge eating. Each item is assessed based on 1 of 4 responses, with 1 denoting that a participant has greater control over eating behavior and 4 denoting that a participant had less control over eating behavior. A total score (sum of the 16 items) may range from 16-64. A lower score indicates greater control over eating behavior.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 184 | 189
units on a scale | -8.55 (0.763) | -18.87 (0.755)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures Analysis — Multiplicity is not adjusted for this secondary efficacy endpoint in this study; Least squares mean difference = -10.32, 95% CI 2-sided [-12.43 to -8.21]

13. Secondary Outcome: Change From Baseline in Frontal Systems Behavior (FrSBe) Total Score at Week 12
Description: The FrSBe is a 46-item self-rating scale designed to measure the neurobehavioral traits associated with the 3 primary regions of the prefrontal cortex. Participants were asked to indicate the frequency with which they have engaged in certain behaviors using a rating scale from "1" (almost never) to "5" (almost always). Summary scores were calculated and converted to t-score. A decrease from baseline in FrSBe total score represents improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: t-scores
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 182 | 187
t-scores | -3.09 (0.592) | -3.40 (0.572)
Statistical Analysis 1: Comparison: PLACEBO vs SPD489; Test type: Superiority or Other; p = 0.706, ANCOVA — Multiplicity is not adjusted for this secondary efficacy endpoint in this study; Least squares mean difference = -0.31, 95% CI 2-sided [-1.93 to 1.31]

14. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self-Report (EQ-5D-5L): Mobility
Description: Quality of life was assessed using the EQ-5D-5L, which is one of the most widely used generic index measures of health-related quality of life. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Percentage of participants with various mobility conditions were reported.
Time Frame: Up to 12 weeks
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 178 | 187
percentage of participants
  No problems walking about | 82.6 | 87.2
  Slight problems walking about | 14.0 | 10.7
  Moderate problems walking about | 2.8 | 2.1
  Severe problems walking about | 0.6 | 0
  Unable to walk about | 0 | 0

15. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self-Report (EQ-5D-5L): Self-Care
Description: Quality of life was assessed using the EQ-5D-5L, which is one of the most widely used generic index measures of health-related quality of life. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Percentage of participants with various self-care conditions were reported.
Time Frame: Up to 12 weeks
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 178 | 187
percentage of participants
  No problems washing or dressing | 89.3 | 95.7
  Slight problems washing or dressing | 6.7 | 3.2
  Moderate problems washing or dressing | 3.9 | 1.1
  Severe problems washing or dressing | 0 | 0
  Unable to wash or dress | 0 | 0

16. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self-Report (EQ-5D-5L): Usual Activities
Description: Quality of life was assessed using the EQ-5D-5L, which is one of the most widely used generic index measures of health-related quality of life. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Percentage of participants with various usual activities conditions were reported.
Time Frame: Up to 12 weeks
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 177 | 186
percentage of participants
  No problems doing usual activities | 78.0 | 87.1
  Slight problems doing usual activities | 14.7 | 9.7
  Moderate problems doing usual activities | 6.2 | 3.2
  Severe problems doing usual activities | 1.1 | 0
  Unable to do usual activities | 0 | 0

17. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self-Report (EQ-5D-5L): Pain/Discomfort
Description: Quality of life was assessed using the EQ-5D-5L, which is one of the most widely used generic index measures of health-related quality of life. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Percentage of participants with various pain/discomfort conditions were reported.
Time Frame: Up to 12 weeks
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 178 | 187
percentage of participants
  No pain or discomfort | 64.6 | 71.1
  Slight pain or discomfort | 27.5 | 20.9
  Moderate pain or discomfort | 7.3 | 7.5
  Severe pain or discomfort | 0.6 | 0.5
  Extreme pain or discomfort | 0 | 0

18. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self-Report (EQ-5D-5L): Anxiety/Depression
Description: Quality of life was assessed using the EQ-5D-5L, which is one of the most widely used generic index measures of health-related quality of life. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Percentage of participants with various anxiety/depression conditions were reported.
Time Frame: Up to 12 weeks
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 178 | 187
percentage of participants
  Not anxious or depressed | 70.2 | 72.2
  Slightly anxious or depressed | 19.7 | 16.6
  Moderately anxious or depressed | 7.9 | 9.1
  Severely anxious or depressed | 2.2 | 1.6
  Extremely anxious or depressed | 0 | 0.5

19. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a semi-structured interview that captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behaviour occurred. The assessment is done by the nature of the responses, not by a numbered scale. Number of participants with suicidal ideation and suicidal behavior were reported.
Time Frame: Up to 12 weeks
Population: The Safety Analysis Set was defined as all randomized participants who took at least 1 dose of investigational product and who had at least 1 post-baseline safety assessment completed. Not all participants had data for this outcome.
Measure: Number; unit: participants
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 187 | 191
participants
  Suicidal Ideation | 3 | 2
  Suicidal behavior | 0 | 0

20. Secondary Outcome: Amphetamine Cessation Symptom Assessment (ACSA) Total Score
Description: ACSA scale has 16 symptom items rated on a scale from 0 (not at all) to 4 (extremely) with a possible total score range of 0 to 64. Higher scores indicate greater withdrawal symptom severity.
Time Frame: Up to 12 weeks
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PLACEBO | SPD489
Number analyzed (Participants) | 138 | 155
units on a scale | 7.3 (7.74) | 5.7 (7.37)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 3 days after the last dose at up to 12 weeks
Arm/Group | PLACEBO | SPD489
Serious Adverse Events (participants affected / at risk) | 2/187 | 3/192
Other Adverse Events (participants affected / at risk) | 67/187 | 125/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=187) | SPD489 (N=192)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=187) | SPD489 (N=192)
Constipation (Gastrointestinal disorders) | 4 (4) | 11 (11)
Dry mouth (Gastrointestinal disorders) | 16 (19) | 76 (86)
Nausea (Gastrointestinal disorders) | 14 (15) | 16 (19)
Fatigue (General disorders) | 10 (11) | 7 (7)
Feeling jittery (General disorders) | 2 (3) | 11 (13)
Irritability (General disorders) | 13 (13) | 16 (18)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 8 (10)
Heart rate increased (Investigations) | 5 (5) | 14 (14)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 17 (17)
Headache (Nervous system disorders) | 17 (19) | 26 (32)
Anxiety (Psychiatric disorders) | 2 (2) | 13 (13)
Insomnia (Psychiatric disorders) | 14 (15) | 34 (44)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.